CLINICAL TRIAL: NCT02713308
Title: Impact of MultiPoint Pacing Technology in CRT Patients With Reduced RV-to-LV Delay
Acronym: IMAGE-CRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Monaldi Hospital (Other)
Responsible Party: Principal Investigator, Antonio D'Onofrio, MD, Monaldi Hospital
Other Study IDs: MP001
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group1-CRT: Patients with RV-to-LV delay≥80ms, CRT standard programming (single-point)
- Group2-MPP: Patients with RV-to-LV delay<80ms, CRT programming with MPP (multi-point)

SUMMARY:
Observational, retrospective and perspective study with acute and chronic endpoints

DETAILED DESCRIPTION:
Study to assess the benefit from Multipoint Pacing (MPP) in presence of RV-to-LV delay<80ms in terms of rate of CRT responder patients at 6 Months from CRT-D system implantation

ELIGIBILITY:
Inclusion Criteria:

* Indication to CRT-D system implantation according to current guidelines or CRT-D system already implanted in patient scheduled to CRT-D system implantation according to current guidelines

Exclusion Criteria:

* Right Bundle Branch Block
* Severe Irreversible Renal Failure (eGFR<30)
* NYHA IV
* Atrio-Ventricular Block above the 1st grade
* Prosthetic Valves
* Atrial Fibrillation at implantation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with standard indication to CRT-D system implantation
Sampling Method: Probability Sample
Enrollment: 248 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Rate of CRT responder patients | 6 Months
  A patient is considered "responder" if Left Ventricular End-Systolic Volume at 6 Months from CRT-D system implantation is reduced at least of 15% towards the baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Antonio D'Onofrio, MD, Study Chair — Monaldi Hospital
Locations (2):
- Italy (2):
  - Monaldi Hospital, Naples
  - Università della Campania "Luigi Vanvitelli", Naples

REFERENCES:
- [Derived] Solimene F, Nigro G, Canciello M, Tavoletta V, Shopova G, Calvanese R, Rago A, La Rosa C, Nappi F, Viscusi M, Urraro F, Manzo G, Gallo P, Andriani A, Rovaris G, Palmisano P, Innocenti S, D'Onofrio A. Design and rationale of the Impact of MultiPoint pacing in CRT patients with reduced RV-to-LV delay (IMAGE-CRT) study. J Cardiovasc Med (Hagerstown). 2020 Mar;21(3):250-258. doi: 10.2459/JCM.0000000000000928. PMID 32004245